CLINICAL TRIAL: NCT04030169
Title: An Open-Label, Phase 2, Multicenter Feasibility Study of Manualized MDMA-Assisted Psychotherapy With an Optional fMRI Sub-Study Assessing Changes in Brain Activity in Subjects With Posttraumatic Stress Disorder
Brief Title: Open Label Study of MDMA-assisted Psychotherapy for Treatment of PTSD With Optional fMRI Sub-Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MAPS Europe B.V. (Industry)
Collaborators: Multidisciplinary Association for Psychedelic Studies (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MP18
Record Dates: First submitted 2019-07-19; First posted 2019-07-23 (Actual); Results first posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: PTSD
Keywords: MDMA; methylenedioxymethamphetamine; psychotherapy; PTSD; Posttraumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — N-Methyl-3,4-methylenedioxyamphetamine

STUDY DESIGN:
Intervention Model Description: Examining safety and effects of two sessions of MDMA-assisted psychotherapy, with Clinician-Administered PTSD Scale for DSM 5 (CAPS-5) severity after treatment compared with baseline
Masking Description: This study will be open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Experimental: MDMA-assisted psychotherapy (Experimental): Administration of 80 to 120 mg midomafetamine (MDMA) HCl followed by a supplemental half-dose 1.5 to 2 hrs after the initial dose of 40 or 60 mg, respectively, in combination with manualized psychotherapy.
  Interventions: Drug: Midomafetamine HCl

INTERVENTIONS:
Drug: Midomafetamine HCl — Non-directive psychotherapy conducted during MDMA-assisted psychotherapy session
  Other Names: 3,4-methylenedioxymethamphetamine; MDMA; MDMA HCl; Midomafetamine

SUMMARY:
The goal of this clinical trial is to learn if MDMA-assisted therapy is safe and effective in people diagnosed with at least severe PTSD.

The main question it aims to answer is: Do two open-label sessions of MDMA-assisted therapy reduce PTSD symptoms?

Participants will receive three non-drug preparatory sessions followed by two sessions of MDMA-assisted therapy. Each MDMA-assisted therapy session is followed by three non-drug integrative therapy sessions.

DETAILED DESCRIPTION:
This multi-site, open-label, Phase 2, lead-in study conducted in Europe assesses the safety and efficacy of MDMA-assisted therapy in participants diagnosed with at least severe posttraumatic stress disorder (PTSD). This study additionally provides an opportunity for clinical supervision to planned Phase 3 therapy teams. Select sites will also participate in an optional fMRI (brain imaging) sub-study.

This study compares the effects of two open-label manualized Experimental Sessions of psychotherapy assisted by flexible doses of MDMA HCl. Initial doses per Experimental Session include 80 mg or 120 mg of MDMA HCl, followed 1.5 to 2 hours later by a supplemental half-dose (40 mg or 60 mg). Total amounts of MDMA to be administered per Experimental Session range from 80 mg to 180 mg. This ~8-week Treatment Period is preceded by three non-drug Preparatory Sessions. During the Treatment Period, each Experimental Session is followed by three Integrative Sessions of non-drug psychotherapy.

The primary endpoint is the change in Clinician Administered PTSD Scale for DSM 5 (CAPS-5) from Baseline to 13 weeks post-baseline (Visit 14). The secondary endpoint is the change in Sheehan Disability Scale (adapted SDS) item scores from Baseline to 13 weeks post-baseline (Visit 14).

ELIGIBILITY:
Inclusion Criteria:

1. Are at least 18 years old
2. Are fluent in speaking and reading the predominantly used or recognized language of the study site
3. Are able to swallow pills
4. Agree to have study visits video-recorded, including Experimental Sessions, Independent Rater assessments, and non-drug psychotherapy sessions
5. Must provide a contact (relative, spouse, close friend or other support person) who is willing and able to be reached by the investigators in the event of a participant becoming suicidal or unreachable
6. Must agree to inform the investigators within 48 hours of any medical treatments and procedures
7. People able to become pregnant (PABP) (i.e., assigned female at birth, fertile, following menarche and until becoming post-menopausal unless permanently sterile), must have a highly sensitive negative pregnancy test at study entry and prior to each Experimental Session, and must agree to use adequate birth control through 10 days after the last Experimental Session. Adequate birth control methods include intrauterine device (IUD), injected or implanted hormonal methods, abstinence, oral hormones plus a barrier contraception, vasectomized sole partner.
8. Agree to the following lifestyle modifications: comply with requirements for fasting and refraining from certain medications prior to Experimental Sessions, not enroll in any other interventional clinical trials during the duration of the study, remain overnight at the study site after each Experimental Session and be driven home after, and commit to medication dosing, therapy, and study procedures

Exclusion Criteria:

1. Are not able to give adequate informed consent
2. Have any current problem which, in the opinion of the investigator or Medical Monitor, might interfere with participation
3. Would present a serious risk to others as established through clinical interview and contact with treating psychiatrist
4. Require ongoing concomitant therapy with a psychiatric medication (exceptions apply)
5. Weigh less than 48 kilograms (kg)
6. Are pregnant or nursing or are able to become pregnant and are not practicing an effective means of birth control.
7. Have a history of any medical condition that could make receiving a sympathomimetic drug harmful because of increases in blood pressure (BP) and heart rate.
8. Have current alcohol or substance use disorder.
9. Have used Ecstasy (material represented as containing MDMA) more than 10 times within the last 10 years or at least once within 6 months of the first Experimental Session; or have previously participated in a clinical trial conducted by the sponsor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2020-06-24 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2023-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Eric Vermetten, MD, Principal Investigator — Leiden University Medical Center
Locations (6):
- NUDZ - National Institute of Mental Health, Klecany, Central Bohemia, Czechia
- Charité - Universitätsmedizin, Berlin Campus Benjamin Franklin, Berlin, Germany
- Stichting Centrum '45/Arq, Oegstgeest, Noord Holand, Netherlands
- Sykehuset Østfold Hf, DPS Norder, Moss, Norway
- United Kingdom (2):
  - University Hospital of Wales - Research Facility, Cardiff
  - The Institute of Psychiatry, Psychology and Neuroscience, London

IPD SHARING:
Plan to Share IPD: Yes
We will share outcome data appearing in any published reports upn request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data and study-related documents will be available when all participants have completed the study.
Access Criteria: Interested persons should correspond with the central contact for the multi-site study.

RESULTS

PARTICIPANT FLOW:
Groups:
- MDMA-assisted Psychotherapy: Open-label administration of 80 to 120 mg midomafetamine HCl in combination with psychotherapy, followed by a supplemental half-dose of 40 or 60 mg offered 1.5 to 2 hrs after the initial dose, respectively.
Period: Overall Study
Arm/Group | MDMA-assisted Psychotherapy
Started | 21
Completed | 20
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | MDMA-assisted Psychotherapy
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.3 (10.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 20
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Netherlands | 8
  Czechia | 3
  Norway | 2
  United Kingdom | 6
  Germany | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in CAPS-5 Total Severity Score
Description: The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) is a 30-item semi-structured interview assessing PTSD in the past month through diagnostic and symptom severity scores anchored to a DSM-5 defined traumatic event. The CAPS-5 produces a Total Severity Score based on severity of PTSD domains described in the DSM-5, as well as a categorical rating indicating whether a participant meets PTSD diagnostic criteria. CAPS-5 Total Symptom Severity scores range from 0 to 80 with higher values designating greater symptom severity. CAPS-5 assigns PTSD diagnosis as being present or absent.
Time Frame: 13 weeks post-baseline
Population: mITT analysis includes 1 participant who did not complete the primary outcome CAPS-5 assessment.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | MDMA-assisted Psychotherapy
Number analyzed (Participants) | 21
score on a scale | -13.95 [-16.32 to -11.58]

2. Secondary Outcome: Change in Sheehan Disability Scale (SDS) Item Scores
Description: The Sheehan Disability Scale (SDS) is a clinician-rated assessment of functional impairment for PTSD. The SDS is a 3-item scale measuring the severity of disability (i.e., the degree of impairment) in the domains of work, family life/home responsibilities and social/leisure activities. Responses are recorded using an 11-point scale (0 = not at all to 10 = extremely) and 5 verbal tags (not at all, mildly, moderately, markedly, extremely). For participants who are not able to work for reasons unrelated to PTSD, the measure includes an option to skip the work-related impairment item, and the reason was collected. The impact of missing item-level data was mitigated by averaging across the items to obtain a Total Score, rather than a straight sum.
Time Frame: 13 weeks post-baseline
Population: mITT analysis includes 1 participant who did not complete the secondary endpoint SDS assessment.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Groups:
- Experimental: MDMA-assisted Psychotherapy: Administration of 80 to 120 mg midomafetamine (MDMA) HCl in combination with manualized psychotherapy, followed by a supplemental half-dose 1.5 to 2 hrs after the initial dose of 40 or 60 mg, respectively.
  Midomafetamine: Non-directive psychotherapy conducted during MDMA-assisted psychotherapy session
Arm/Group | Experimental: MDMA-assisted Psychotherapy
Number analyzed (Participants) | 21
Score on a scale
  Family Life / Home | -1.18 [-2.14 to -0.22]
  Social / Leisure Activities | -1.45 [-2.32 to -0.58]
  Work / School | -1.45 [-2.36 to -0.53]
  Total Score | -1.30 [-2.17 to -0.43]

ADVERSE EVENTS:
Time Frame: Approximately 8 weeks
Description: Treatment Emergent Adverse Events: Adverse events that occur during the treatment period from the first Experimental Session to the last Integrative Session
Arm/Group | Experimental: MDMA-assisted Psychotherapy
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 2/21
Other Adverse Events (participants affected / at risk) | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: MDMA-assisted Psychotherapy (N=21)
Suicidal ideation (Psychiatric disorders) | 1
Suicidal behavior (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Experimental: MDMA-assisted Psychotherapy (N=21)
Palpitations (Cardiac disorders) | 2
Vision blurred (Eye disorders) | 2
Nausea (Gastrointestinal disorders) | 8
Vomiting (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 4
Feeling cold (General disorders) | 2
Feeling hot (General disorders) | 2
Blood pressure increased (Investigations) | 2
Decreased appetite (Metabolism and nutrition disorders) | 4
Muscle tightness (Musculoskeletal and connective tissue disorders) | 8
Back pain (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Headache (Nervous system disorders) | 15
Dizziness (Nervous system disorders) | 2
Paraesthesia (Nervous system disorders) | 2
Tension headache (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 4
Suicidal ideation (Psychiatric disorders) | 7
Dry mouth (Gastrointestinal disorders) | 2
Emotional disorder (Psychiatric disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-11-22): https://cdn.clinicaltrials.gov/large-docs/69/NCT04030169/Prot_000.pdf
  • Statistical Analysis Plan (2019-09-05): https://cdn.clinicaltrials.gov/large-docs/69/NCT04030169/SAP_001.pdf
  • Informed Consent Form (2022-11-22): https://cdn.clinicaltrials.gov/large-docs/69/NCT04030169/ICF_003.pdf